CLINICAL TRIAL: NCT02586753
Title: A Phase II Study to Compare Paclitaxel or S1 Plus Cisplatin in Concurrent Chemoradiotherapy for Squamous Cell Carcinoma of Esophagus
Brief Title: Paclitaxel or S1 Plus Cisplatin in Concurrent Chemoradiotherapy for Squamous Cell Carcinoma of Esophagus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mianyang Central Hospital (Other)
Responsible Party: Principal Investigator, Feng Gao, Principal Investigator, Mianyang Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MianyangCH001
Record Dates: First submitted 2015-10-19; First posted 2015-10-26 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Cisplatin; Radiotherapy; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel plus Cisplatin with radiotherapy (Experimental): patients will receive concurrent chemoradiotherapy with drug Paclitaxel plus Cisplatin
  Interventions: Other: Paclitaxel plus Cisplatin with radiotherapy
- S1 plus Cisplatin with radiotherapy (Experimental): patients will receive concurrent chemoradiotherapy with drug S1 plus Cisplatin
  Interventions: Other: S1 plus Cisplatin with radiotherapy

INTERVENTIONS:
Other: Paclitaxel plus Cisplatin with radiotherapy — we want to compare which regime is better with radiotherapy, PT regime (paclitaxel and cisplatine ) Chemotherapy: Patients will be concurrently administered with irradiation every 3 weeks with PT regimen (cisplatin of 20 mg/m2/d, d1-3; PTX(paclitaxel)of 135mg/m2/d, d1) for 4 cycles. For the first 2-cycles of chemotherapy they will be concurrently given with irradiation and the remained 2 cycles, after irradiation.
  Radiotherapy:Patients will be conducted CT simulation, and Intensity-modulated radiation therapy(IMRT)was performed. 1.8-2.0 Gy/fraction, 5 fractions a week, with a total dose of 60-66Gy will be delivered for all patients by 6-MV-X-ray of linear accelerator.
  Arms: Paclitaxel plus Cisplatin with radiotherapy
Other: S1 plus Cisplatin with radiotherapy — we want to compare which regime is better with radiotherapy,SP regime (Tegafur Gimeracil Oteracil Potassium Capsule and cisplatine).
  Chemotherapy: Patients will be concurrently administered with irradiation every 3 weeks with PS regimen (cisplatin of 20 mg/m2/d, d1-3; S1(Tegafur Gimeracil Oteracil Potassium Capsule)of 50mg/m2/d, d1-14) for 4 cycles. For the first 2-cycles of chemotherapy they will be concurrently given with irradiation and the remained 2 cycles, after irradiation.
  Radiotherapy:Patients will be conducted CT simulation, and Intensity-modulated radiation therapy(IMRT)was performed. 1.8-2.0 Gy/fraction, 5 fractions a week, with a total dose of 60-66Gy will be delivered for all patients by 6-MV-X-ray of linear accelerator.
  Arms: S1 plus Cisplatin with radiotherapy

SUMMARY:
The purpose of this study is to determine which regimen is better for esophageal squamous carcinoma in concurrent chemoradiation(CCRT),paclitaxel or S1 plus cisplatin.

DETAILED DESCRIPTION:
Radiotherapy:Patients will be conducted CT simulation, and three-dimensional conformal radiation therapy (3DCRT) was performed. 1.8-2.0 Gy/fraction, 5 fractions a week, with a total dose of 60-66Gy will be delivered for all patients by 6-MV-X-ray of linear accelerator.

Chemotherapy: Patients will be concurrently administered with irradiation every 3 weeks with PT regimen (cisplatin of 20 mg/m2/d, d1-3; PTX(paclitaxel)of 135mg/m2/d, d1) for 4 cycles or PS regimen (cisplatin of 20 mg/m2/d, d1-3; S1(Tegafur Gimeracil Oteracil Potassium Capsule)of 50mg/m2/d, d1-14) for 4 cycles. For the first 2-cycles of chemotherapy they will be concurrently given with irradiation and the remained 2 cycles, after irradiation.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven squamous cell carcinoma of esophagus .
2. Locally advanced esophageal cancer , with no operation indication
3. M1a disease defined ( AJCC 1998) , including celiac lymph node for lower thoracic esophageal cancer and cervical lymph node involvement for upper thoracic esophageal cancer
4. Subjects haven't been given neither radiotherapy nor chemotherapy before
5. Age of 18-70
6. PS ≦2
7. Hemogram : WBC≧ 4000/mm3 or ANC ≧ 2000 /mm3 and Platelet ≧ 100,000/mm3 . Biochemistry : GOT/GPT ≦ 3.5 times , Cr ≦ 1.5 mg/dl and Bilirubin ≦ 2.0 mg/dl
8. With no difficulty in eating
9. Expected lifetime ≧3 months

Exclusion Criteria:

1. Invasion to surrounding organ ( T4 disease ) .
2. Distant metastasis , except M1a disease .
3. Complete obstruction of the esophagus, or patients who have the potential to develop perforation
4. Women in status of pregnancy
5. Patients who have complications exist as following:

   * Uncontrolled angina and heart failure, have a history of hospitalization in 3 months
   * A history of myocardial infarction in the past 6 months
   * There is a need for antibiotic treatment of acute bacterial or fungal infection
   * Chronic obstructive pulmonary disease, or other lung disease requiring hospitalization
   * Drug addiction, alcoholism and AIDS disease or long-term virus carriers
   * Uncontrollable seizures, or loss of insight because of mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | five years after enrollment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | five years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Bo X Du, Doctor, Principal Investigator — Mianyang Central Hospital

REFERENCES:
- [Background] Conroy T, Yataghene Y, Etienne PL, Michel P, Senellart H, Raoul JL, Mineur L, Rives M, Mirabel X, Lamezec B, Rio E, Le Prise E, Peiffert D, Adenis A. Phase II randomised trial of chemoradiotherapy with FOLFOX4 or cisplatin plus fluorouracil in oesophageal cancer. Br J Cancer. 2010 Oct 26;103(9):1349-55. doi: 10.1038/sj.bjc.6605943. Epub 2010 Oct 12. PMID 20940718
- See also: Click here for more information about this study: Phase II randomised trial of chemoradiotherapy with FOLFOX4 or cisplatin plus fluorouracil in oesophageal cancer — http://www.bjcancer.com